CLINICAL TRIAL: NCT06713356
Title: Ultrasonographic Assessment in Comparison to MRI in Diagnosis of TMJ Internal Derangement
Brief Title: US Vs MRI in Diagnosis of TMJ Internal Derangement
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Anwar Kamal El Dein Hussien, Resident Doctor, Assiut University
Other Study IDs: TMJ internal derangement
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: TMJ Internal Derangement
Keywords: MRI; US; TMJ; internal derangement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compare the accuracy of ultrasonography and magnetic resonance imaging in the diagnosis of temporomandibular joint internal derangements.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMDs) are conditions that affect the temporomandibular joint (TMJ), often leading to pain and dysfunction. The most common cause of TMJ problems is internal derangements.

The term "internal derangements" refers to conditions with the articular disc displaced from its original position on the mandibular condyle.

Disc displacement may occur anteriorly, anterolaterally, laterally, anteromedially, medially, or posteriorly, but the latter is very rare.

Anterior disc displacement (ADD) is the most common ID condition and is usually divided into two categories: with reduction and without reduction. Each category has special features during closed and opened mouth positions. Therefore, the examination should include both positions.

Clinical examination alone isn't enough to diagnose TMJ problems, therefore additional imaging tests are often needed.

Magnetic resonance imaging (MRI) is the gold standard modality, however because of its limited availability, long scan time, and high cost, it is difficult to use MRI as a screening technique.

Ultrasound (US) has been recommended as an alternate diagnostic imaging modality for TMJ problems as it is less costly, non-invasive and capable of providing real-time imaging, presents an alternative diagnostic tool. Thus, the articular disc may be seen as the patient is opening and closing their mouth

ELIGIBILITY:
Inclusion Criteria:

* Patients showing signs of TMJ internal derangements

Exclusion Criteria:

* contraindications for MRI such as claustrophobia, heart pacemaker and metallic foreign body carriers.
* patients in which the misaligned images or distortions due to motion artifacts made the interpretation of the MRI unreliable.
* Previously operated TMJ.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients showing signs of TMJ internal derangements
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between US and MRI in diagnosis of TMJ disc displacement. | Baseline
  Compare the accuracy of assessment of disc positioning by ultrasonography and magnetic resonance imaging in patients with TMJ disorders
  .

CONTACTS AND LOCATIONS:
Overall Officials: Sami A. Sayed, Study Director — Professor doctor; Omran K. Qenawy, Study Director — Assistant professor doctor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Emshoff R, Kriwanek S, Koller M, et al. Diagnostic accuracy of ultrasound in the assessment of the temporomandibular joint: a comparison with MRI. Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology, and Endodontics. 2022; 96(6):750-756.
- [Result] Salamah T, Harefa GN. Diagnostic value and clinical significance of high-resolution ultrasonography compared to magnetic resonance imaging in diagnosing temporomandibular joint dislocation: a systematic review. Medical Journal of Indonesia. 2024 Mar; 33(1): 29-34.
- [Result] Refaat MM, Yousef MI, Torky AA, Sarow ML. Ultrasonography compared to magnetic resonance imaging for the diagnosis of the temporomandibular joint disc displacement: Benha Journal of Applied Sciences. 2021 Nov; 6(6): 133-43.
- [Result] Li C, Zhou J, Shi Y, Ye Z, Zhang C, Hou R, Li Z, You M. Diagnostic efficacy of quantitative ultrasonography for anterior disc displacement of the temporomandibular joint. Quant Imaging Med Surg. 2023 Oct 1;13(10):6446-6455. doi: 10.21037/qims-23-401. Epub 2023 Aug 3. PMID 37869327
- [Result] Minervini G, Nucci L, Lanza A, Femiano F, Contaldo M, Grassia V. Temporomandibular disc displacement with reduction treated with anterior repositioning splint: a 2-year clinical and magnetic resonance imaging (MRI) follow-up. J Biol Regul Homeost Agents. 2020 Jan-Feb;34(1 Suppl. 1):151-160. DENTAL SUPPLEMENT. PMID 32064850
- [Result] Talmaceanu D, Lenghel LM, Bolog N, Buduru S, Leucuta D, Rotar H. High-resolution ultrasound imaging compared to magnetic resonance imaging for temporomandibular joint disorders: An in vivo study. Eur J Radiol. 2020 Nov;132:109291. doi: 10.1016/j.ejrad.2020.109291. Epub 2020 Sep 17. PMID 32980724
- [Result] Moturi K. Internal derangements of temporomandibular joint. Temporomandibular Joint Disorders: Principles and Current Practice. 2021;: 189-207.
- [Result] Palmer J, Durham J. Temporomandibular disorders. BJA Educ. 2021 Feb;21(2):44-50. doi: 10.1016/j.bjae.2020.11.001. Epub 2020 Dec 24. No abstract available. PMID 33889429